CLINICAL TRIAL: NCT01618045
Title: Nutritional Regulation Of Wound Inflammation: Part II
Acronym: FPPT2DM-II
Status: Completed | Type: Observational
Sponsor: Ohio State University (Other)
Collaborators: Osato Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 20120293
Record Dates: First submitted 2012-06-11; First posted 2012-06-13 (Estimated); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Diabetes
Keywords: Diabetes; FPP; fermented papaya preparation
MeSH Terms: conditions — Diabetes Mellitus | interventions — fermented papaya preparation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — Blood will be drawn for the study.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Fermented Papaya Preparation (FPP): This a is single arm study - all participants will receive and take fermented papaya preparation (FPP) for a total of 6 weeks. Participants will take 3 grams of FPP three times per day (a total of 9 grams per day).
  Interventions: Dietary Supplement: Fermented Papaya Preparation (FPP)

INTERVENTIONS:
Dietary Supplement: Fermented Papaya Preparation (FPP) — Participants will take fermented papaya preparation (FPP) for a total of 6 weeks (3 grams, three times each day for a total of 9 grams per day). The participants will attend 5 study visits and have their blood draw at each visit (5 total times).
  Other Names: Immun'Age; FPP

SUMMARY:
Fermented Papaya Preparation (FPP) is a sweet and granular substance available over the counter. FPP possesses antioxidant properties, which provide benefit against age-related complications, and is also known to protect red blood cells (RBCs) against oxidative damage and to help protect against severe forms of thalassemia. The investigators recently showed that ex vivo supplementation of FPP can correct respiratory burst performance of diabetic peripheral blood mononuclear cells (PBMC) via a Sp-1 dependant pathway. Based on these observations, the investigators propose to study the outcome that FPP supplementation has in patients with diabetes.

DETAILED DESCRIPTION:
Fermented Papaya Preparation (FPP) possesses antioxidant properties, which provide benefit against age-related complications. FPP is also known to protect red blood cells (RBCs) against oxidative damage and to help protect against severe forms of thalassemia. Several independent observations convergently point toward the hypothesis that treatment with papaya preparations may facilitate wound healing responses. Chronic wounds in patients with diabetes represent a major public health problem. Previous studies from the investigators have demonstrated that wound-site macrophages from patients with diabetes are compromised in their ability to support wound healing. Recently, our laboratory reported the first evidence demonstrating that FPP may improve diabetic wound outcomes by specifically influencing the response of wound-site macrophages and the subsequent angiogenic response. FPP has a long track record of safe human consumption.

The objective of the current study is to determine whether FPP is able to improve inducible respiratory burst outcomes in peripheral blood mononuclear cells (PBMC) of participants with diabetes. Our investigators have recently reported that supplementation with standardized fermented papaya preparation (FPP) in adult diabetic mice improves dermal wound healing outcomes. The production of reactive oxygen species (ROS) by type 2 diabetics (T2DM) PBMC is markedly inhibited compared to that of the PBMC from non-diabetic donors. We observed that ex vivo FPP supplementation corrected such inhibition in ROS production by PBMC from T2DM donors. Therefore, based on these observations, the investigators propose to study the outcome that FPP supplementation has in patients with diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients 30 to 80 years old with clinically defined type II diabetes and HbA1c ≤ 9.0 and BMI between 22 and 42
* Diabetic subjects selected for the study will meet one or more of the following criteria as recommended by American Diabetes Association:
* 1) Symptoms of diabetes and casual plasma glucose 200 mg/dl (11.1 mmol/l) (casual is defined as any time of day without regard to time since last meal. The classic symptoms of diabetes include polyuria, polydipsia, and unexplained weight loss); OR
* 2) Fasting plasma glucose (FPG) 126 mg/dl (7.0 mmol/l) (fasting is defined as no caloric intake for at least 8 h); OR
* 3) 2-hr plasma glucose 200 mg/dl (11.1 mmol/l) during an oral glucose tolerance test (OGTT) (this test should be performed as described by the World Health Organization, using a glucose load containing the equivalent of 75g anhydrous glucose dissolved in water)

Exclusion Criteria:

* Individuals who are deemed unable to understand the procedures, risks and benefits of the study (i.e., informed consent) will be excluded
* T2DM with HbA1c = 9.1 or above
* BMI less than 22 and over 42
* Clinically significant kidney or liver disease
* Severe neurologic dysfunction
* Females who are pregnant as well as individuals who are therapeutically immuno-compromised will also be excluded in order to minimize the risk to such individuals (and fetus) and to decrease statistical variability and to minimize the potential of confounders
* Candidates for inclusion into the study will not include individuals as defined in 45 CFR 46 Subparts B, C and D, nor from any other population which may be considered vulnerable
* Pregnant women are excluded to minimize the risk to such individuals (and fetus) and to decrease statistical variability and to minimize the potential of confounders

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The subject population in this study will be patients with type 2 diabetes with the following parameters.
  * Age 30 to 80 years old
  * HbA1c ≤ 9. 0
  * BMI between 22-42
Sampling Method: Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2012-05; Primary Completion 2015-01-19 (Actual); Study Completion 2015-02-19 (Actual)

PRIMARY OUTCOMES:
Blood glucose level | Initial visit, 2 weeks of FPP supplementation, 6 weeks of FPP supplementation, 1 week after stopping FPP supplementation, and 2 weeks after stopping FPP supplementation
  The blood glucose level will be measured from blood drawn via venipuncture at each study visit throughout the duration of the study.
HbA1c level | Initial visit, 2 weeks of FPP supplementation, 6 weeks of FPP supplementation, and 2 weeks after stopping FPP supplementation
  HbA1c level will be measured from blood drawn from venipuncture to assess any change in the level during FPP supplementation and after stopping FPP supplementation.
Monocyte Function | Initial visit, 2 weeks of FPP supplementation, 6 weeks of FPP supplementation, 1 week after stopping FPP supplementation, and 2 weeks after stopping FPP supplementation
  Blood drawn from venipuncture at each study visit will be assessed to determine monocyte reactive oxygen species (ROS) production and NADPH oxidase expression (Rac2 levels).

SECONDARY OUTCOMES:
Lipid Profile | Initial visit, 6 weeks of FPP supplementation, and 2 weeks after stopping FPP supplementation
  Lipid profile (cholesterol levels) will be measured from blood drawn via venipuncture to assess for any changes during FPP supplementation and after stopping FPP supplementation.

CONTACTS AND LOCATIONS:
Overall Officials: Sashwati Roy, PhD., Principal Investigator — Ohio State University
Locations (5):
- United States (5):
  - OSU CarePoint East, Columbus, Ohio
  - University Hospital East (Wound Center), Columbus, Ohio
  - University Hospital East, OSUWMC Diabetes Clinic, Columbus, Ohio
  - The Ohio State University/Ohio State University Wexner Medical Center, Columbus, Ohio
  - OSUWMC Comprehensive Wound Care Center, Martha Morehouse Medical Plaza, Columbus, Ohio